CLINICAL TRIAL: NCT05434819
Title: Surgical Ablation of AF Efficacy Trial
Acronym: SAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Richard Whitlock, Professor of Surgery, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAFEV1.0
Record Dates: First submitted 2022-05-04; First posted 2022-06-28 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Surgical Ablation; Cardiac Surgery
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Intervention Model Description: Each patient will be assigned in a blinded fashion to one of two groups (atrial fibrillation ablation or no atrial fibrillation ablation) in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding to allocation will be maintained for all parties, excluding the operating surgeon and necessary operating room personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Atrial Fibrillation Ablation Group (Experimental): Surgeon will perform left atrial ablation during patient's cardiac surgery procedure.
  Interventions: Procedure: Surgical Atrial Fibrillation Ablation
- No Surgical Atrial Fibrillation Ablation Group (No Intervention): Surgeon will not perform left atrial ablation during the patient's cardiac surgery procedure.

INTERVENTIONS:
Procedure: Surgical Atrial Fibrillation Ablation — Surgeon will preform surgical atrial fibrillation ablation using either cryoablation or bipolar radiofrequency clamps including 2 layers of atrium or vein, a minimum of 2 burns per clamping with at least 3 lines in the ablation group. Cavo-tricuspid isthmus and mitral lines will be allowed.
  Arms: Surgical Atrial Fibrillation Ablation Group

SUMMARY:
SAFE is an international multicentre RCT of concomitant surgical atrial fibrillation (AF) ablation in patients with paroxysmal or persistent AF undergoing cardiac surgery.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) affects more than 1% of the general population and is an important risk factor for stroke. AF prevalence increases with age, occurring in 10 to 15% of patients older than 80 years of age, which is important with the aging population. Of patients undergoing cardiac surgery, 10.8% have a history of AF. AF is believed to cause the left atrium to dilate and lose its transport function. AF significantly increases the risk of ischemic stroke of cardioembolic origin, but is also associated with heart failure and impairs quality of life. Although the causal relationship between the 2 clinical entities has not been fully elucidated, AF is believed to cause heart failure via several mechanisms.

Ablation of AF is the application of scars to the atrial tissue to disrupt faulty electrical signals that cause the arrhythmia. If surgical ablation of AF yields a benefit similar to catheter-based AF ablation, thousands of people undergoing cardiac surgery could benefit from this procedure each year. SAFE will be a landmark trial in cardiac surgery, definitely establishing surgical AF ablation's impact on cardiovascular outcomes. Cardiac surgery is the optimal setting to establish whether maintenance of sinus rhythm through AF ablation yields clinical benefit, and is a setting where sham-control is possible. This will not only provide evidence for the cardiac surgical patients but will bolster the evidence for ablation (catheter or stand-alone surgical) in other AF patients.

The intervention under investigation is concomitant surgical AF ablation which is compared to no surgical AF ablation. The primary outcome is hospital readmissions with heart failure during 4 years of follow-up. This study will enroll 2000 patients from 50 centres, globally. Patients will be followed at hospital discharge, 4 to 6 weeks after surgery, 6 months after surgery, and then at 6-month intervals until the final follow-up visit, for a median follow-up for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Undergoing a clinically indicated cardiac surgical procedure: CABG, AVR, ascending aorta replacement, or combinations thereof;
* Documented history of paroxysmal or persistent AF
* Provide informed consent

Exclusion Criteria:

* Dominant atrial arrhythmia is atrial flutter;
* Documented left atrial diameter ≥ 6 cm;
* Previous cardiac surgery requiring opening of the pericardium;
* Patients undergoing any of the following procedures:

  1. Heart transplant
  2. Complex congenital heart surgery
  3. Sole indication for surgery is ventricular assist device insertion
  4. Mitral valve repair or replacement
  5. Tricuspid valve repair or replacement
* Patient resides in a long-term care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of hospital readmissions for heart failure over duration of follow-up | Common termination point for trial (median follow-up of 4 years)
  Total number of hospital readmissions for heart failure.

SECONDARY OUTCOMES:
Number of Ischemic stroke or systemic arterial embolism events over duration of follow up | Common termination point for trial (median follow-up of 4 years)
  Number of Ischemic stroke or systemic arterial embolism events over duration of follow up
Length of ICU stay | From the date of study intervention surgery completion to the date of index hospital discharge, assessed up to the common termination point for trial (median follow-up of 4 years)
  Length of ICU stay, including readmissions, from study intervention surgery to hospital discharge, including readmissions
Length of hospital stay | From the date of study intervention surgery completion to the date of index hospital discharge, assessed up to the common termination point for trial (median follow-up of 4 years)
  Length of hospital stay
Freedom from recurrence of atrial tachyarrhythmia | 1 year post-operatively
  Freedom from recurrence of atrial tachyarrhythmia
Number of days free from admission to healthcare facility or presentation to the emergency department for heart failure | Common termination point for trial (median follow-up of 4 years)
  Number of days free admission to healthcare facility or presentation to the emergency department for heart failure
All-cause mortality | Common termination point for trial (median follow-up of 4 years)
  All-cause mortality
Cardiovascular mortality | Common termination point for trial (median follow-up of 4 years)
  Cardiovascular mortality
Antiarrhythmic drug use | Beyond 6 weeks until common termination point for trial (median follow-up of 4 years)
  Antiarrhythmic drug use
Number of patients undergoing atrial fibrillation ablation | 90 days post- study surgery until common termination point for trial (median follow-up of 4 years)
  Number of patients undergoing atrial fibrillation ablation
Quality of Life - atrial fibrillation specific | At 1 year, and at common termination point for trial (median follow-up of 4 years)
  Atrial fibrillation specific quality of life as assessed by the Atrial Fibrillation Effect on QualiTy of Life questionnaire (AFEQT) which is 20 questions using a 7 point Likert scale where a higher score means a worse outcome.
Quality of Life - heart failure specific | At 1 year, and at common termination point for trial (median follow-up of 4 years)
  Heart failure specific quality of life assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) which is a 12 questions using Likert scales where a higher score is a better outcome.
Quality of Life - General | At 1 year, and at common termination point for trial (median follow-up of 4 years)
  Quality of life- general as assessed by the European quality of life index version 5D (EQ-5D-5L) which consists of a descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

OTHER OUTCOMES:
Number of Ischemic stroke and systemic arterial embolism | Up to 30 days post-operatively
  Safety outcome
Number of patients requiring permanent pacemaker implantation | Up to 1 year post-operatively
  Safety outcome
Volume of chest tube output | Up to 24 hours post-operatively
  Safety outcome - chest tube output measured in mL.
Re-operation for bleeding | From date of study intervention surgery completion to date of index hospital discharge, assessed up to the common termination point for trial (median follow-up of 4 years)
  Safety outcome
All-cause mortality | Prior to discharge or within 30 days post-operatively (whichever occurs first)
  Safety outcome
Post-operative major bleeding | <48 hours after surgery
  Safety outcome
Number of patients with pulmonary vein stenosis | At 1 year, and at common termination point for trial (median follow-up of 4 years)
  Safety outcome
Number of patients with stiff left atrium syndrome | At 1 year, and at common termination point for trial (median follow-up of 4 years)
  Safety outcome
Number of patients with esophageal to atrial fistula | At 1 year, and at common termination point for trial (median follow-up of 4 years)
  Safety outcome
Health economic analysis of surgical atrial fibrillation | At 1 year, and at common termination point (median follow-up of 4 years)
  Economic analysis will be assessed via health care utilization by patients
Health economic analysis of surgical atrial fibrillation | At 1 year, and at common termination point (median follow-up of 4 years)
  Economic analysis will be assessed via a questionnaire of health care visits and costs incurred by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, Principal Investigator — Population Health Research Institute; Emilie Belley-Côté, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada